CLINICAL TRIAL: NCT04523415
Title: The Reliability and Reproducibility of Edelson Classification About Proxima Humeral Fractures
Brief Title: Researches About Proximal Humerus Fractures
Status: Recruiting | Type: Observational
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JLGuo001
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Proximal Humeral Fracture
Keywords: Proximal Humeral; Fracture; Classifications
MeSH Terms: conditions — Shoulder Fractures; Fractures, Bone | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients wiht CT data: all patients with CT data are enrolled with this research, and the classification about proximal humeral fractures are identified.
  Interventions: Other: without intervention, just retrospectively review the data about patients

INTERVENTIONS:
Other: without intervention, just retrospectively review the data about patients — without intervention

SUMMARY:
Majority of previous classifications based on two-dimensional images to analyze these complicated 3-D fractures. Small or delicate changes in rotation and positioning can result to considerable disagreement in the interpretation of standard radiographs. Therefore, a classification system which had a better reliability and reproducibility for the fractures is warranted and helpful for orthopedic surgeons. Furthermore, CT and 3-D CT construction images with high resolution give a much clearer view of the pattern of proximal humeral fractures. Edelson proposed a new three-dimensional classification for fractures of the proximal humerus. The results concluded that it was a useful in classifying these injuries with reasonable interobserver reliability.

It could be hypothesized that patients with proximal humeral fractures would benefit from this 3D classification, but there is a scarcity of application of the classification in large samples. T

ELIGIBILITY:
Inclusion Criteria:

* Whole imaging data ;
* Clear record of demographic data;
* Three dimensional construction with mimics (with CT of B30);
* Patients older than 17 years with displaced PHF occurring less than 3 weeks before allocation and treatment.

Exclusion Criteria:

* Patients with the presence of neurological disease (syringomyelia and);
* Open fractures;
* Pathological fracture (other than osteoporotic);
* Not a resident in the hospital catchment area

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: proximal humeral fractures without Pathological fracture
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
classification based on Edelson classifications | 2019.01-2022.12

CONTACTS AND LOCATIONS:
Locations (1):
- the Third Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: after the experiment was conducted
Access Criteria: all authors focusing on proximal humeral fractures